CLINICAL TRIAL: NCT04276051
Title: Effects of Vagus Nerve Cryoablation on Glycemic Control and Weight Loss in Obese Patients With Type 2 Diabetes
Brief Title: Cryovagotomy Diabetes Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Alexandra Migdal, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00109624
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Type 2; Diabetes Mellitus; Obesity
Keywords: Obesity; Diabetes; Neurophysiology; Cryovagotomy; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cryoablation of the Vagus Nerve Plus Lifestyle Intervention (Experimental): Participants randomized to receive cryoablation of the vagus nerve as well as standardized dietary and exercise counseling from a registered dietitian and exercise physiologist.
  Interventions: Device: Cryoablation of the Vagus Nerve; Behavioral: Lifestyle Intervention
- Lifestyle Intervention Only (Active Comparator): Participants randomized to receive standardized dietary and exercise counseling from a registered dietitian and exercise physiologist.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Device: Cryoablation of the Vagus Nerve — The Visual ICE Cryoablation System is a mobile console system intended for cryoablative tissue destruction using a minimally invasive procedure. The Visual-ICE System uses high-pressure argon gas that circulates through closed-tip cryoablation needles to induce tissue freezing. Active tissue thawing is achieved by circulating helium gas through the needles or, alternatively, by the use of Galil Medical i-Thaw technology. The procedure will be done under CT guidance and involves a 4-5 mm scalpel incision followed by percutaneous probe placement about the posterior gastroesophageal junction (the location of the posterior vagal trunk). The probe will create a zone of decreased temperature (-20 to -40 degrees Celsius) involving the posterior vagal nerve fibers/plexus. The cryoablation process will include a 3-minute freeze, followed by a 1-minute thaw, and a second 3-minute freeze and 1 minute thaw.
  Other Names: Visual ICE Cryoablation System
  Arms: Cryoablation of the Vagus Nerve Plus Lifestyle Intervention
Behavioral: Lifestyle Intervention — The lifestyle intervention structure will include three face-to-face counseling sessions at baseline, 3 and 6 months. Dietary counseling to follow a low carbohydrate diet will be provided by a registered dietitian. Focus will be on increasing fruits and vegetables and decreasing refined sugars and processed foods. It will also include motivational interviewing, goal setting and nutrition education. In addition, subjects will be encouraged by exercise physiologist to slowly increase physical activity to at least 150 minutes weekly. There will be weekly phone calls or texts (participants' choice) providing a total of 26 points of contact recommended by the United States Preventive Services Task Force.

SUMMARY:
The pilot study will assess the feasibility and efficacy of cryoablation procedure to freeze the vagus nerve in obese patients with type 2 diabetes. Aim 1 will focus on changes in glycemic control. Aim 2 will evaluate differences in body weight and anthropometric measurements. This study will provide much needed data for a novel therapeutic intervention to manage obese patients with type 2 diabetes.

DETAILED DESCRIPTION:
Obesity is a growing epidemic, currently affecting over 1/3 of the adult US population and is a well-established risk factor for the development of diabetes and cardiovascular disease. Given that the majority of patients with type 2 diabetes (T2D) are obese, weight loss is the cornerstone of treatment, and has been shown to decrease risk of long term complications, lead to improvements in A1c and lipid levels, as well as decreased need for medications and improvements in quality of life. Unfortunately, lifestyle intervention is often ineffective at achieving long-term sustainable, clinically significant weight loss. Bariatric surgery is a successful intervention, leading to 20-30% weight loss with remission of diabetes in 30-65% of patients 1-5 years post surgery. However, this invasive procedure is associated with high rates of short- and long-term complications, including need for reoperations, vitamin/mineral deficiencies, anemia, and osteoporosis. It is clear that the current management options for obese patients, including lifestyle changes, medications and surgery, are suboptimal and innovative strategies are necessary to optimize diabetes control and weight management.

Energy balance and glycemic control are mediated largely by the gut-brain axis, specifically the vagus nerve. The vagus nerve can stimulate or inhibit food intake depending on nutritional status. Vagal nerve signaling is disrupted in the setting of obesity and thought to contribute to overeating behaviors. Vagus nerve blockade has the potential to be a highly efficacious, minimally invasive intervention to address current obesity treatment limitations. Clinical studies evaluating the efficacy of an implantable electric vagus nerve blockade device found that subjects lost on average 8.8% of total body weight at 1 year; patients with T2D experienced improved glycemic control, with an average A1c improvement of 1.0% at 12 months. Unfortunately, nearly 40% of subjects experienced side effects related to the device. A recent pilot study from the researchers of this study reported weight loss efficacy of a minimally invasive computerized tomography (CT) guided cryoablation of the vagus nerve in obese, non-diabetic subjects. Patients lost 5.6% of total body weight and 22.7% excess body weight at 6 months with no significant side effects. The purpose of this current study is to evaluate the feasibility and efficacy of this procedure through a randomized control trial in obese patients with T2D. The researchers hypothesize that those patients undergoing the cryoablation procedure will experience improvement in glycemic control and enhanced weight loss at 6 months follow-up compared to the control group.

Participants will be randomized to receive either CT guided cryoablation of the vagus nerve plus lifestyle intervention or lifestyle intervention alone. The lifestyle intervention lasts for 26 weeks and participants will be followed for 12 months in total.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 22-65
2. Diagnosis of type 2 diabetes mellitus (T2DM) for <10 years
3. HbA1c between ≥7.5% and ≤10.5%
4. Treatment with non-insulin antidiabetic medications with stable doses for at least 3 months, with failed prior attempts at dietary interventions to optimize diabetes control
5. BMI 30-40 kg/m^2
6. Willing to comply with study requirements
7. Documented negative pregnancy test in women of child bearing potential and use of an effective birth control method
8. Average score of ≥3 on questions 4, 8, 9, 13, and 14 from the Three Factor Eating Questionnaire

Exclusion Criteria:

1. Diagnosis of type 1 diabetes or history of diabetic ketoacidosis
2. Use of insulin therapy
3. Significant kidney disease (eGFR < 60 ml/min/1.73m^2)
4. Current drug or alcohol addiction
5. Thyroid disease unless underlying diagnosis is primary hypothyroidism on stable medications for >3 months with thyroid stimulating hormone (TSH) in reference range at time of screening visit
6. Systemic steroid use within 30 days prior to randomization
7. Use of prescription or over the counter weight loss medications within 6 months prior to randomization
8. Weight gain/loss >5% over the past 6 months
9. Previous GI surgery or abnormal GI anatomy which may limit technical feasibility of the procedure
10. Recent diagnosis of cardiovascular disease requiring percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) within the past 6 months
11. Abnormal pathologies or conditions of the GI tract, including peptic ulcers, hiatal hernia, active gallbladder disease, pancreatitis, cirrhosis, inflammatory bowel disease, upper GI bleed within 6 months of randomization
12. Any condition or major illness that places the subject at undue risk by participating in the study
13. Psychiatric condition rendering the subject unable to understand the possible consequences of the study
14. Inability to provide informed consent
15. Female subjects who have been pregnant within 6 months or breast-feeding at time of enrollment into the study, or women who plan to become pregnant within the next 12 months
16. Diagnosis of anemia, red blood cell (RBC) transfusion in the preceding 3 months or expectation to receive transfusion within the next 12 months, or hemoglobinopathies that would affect HbA1c reliability
17. Active or recent infection
18. Immunosuppression
19. History of coagulopathy or high risk for development of deep vein thrombosis (including congestive heart failure, those who are non-ambulatory, active leukemia/lymphoma, prior thrombotic events, family history of thrombosis)
20. History of blood pressure instability (systolic BP ≤100 or ≥160 mmHg)
21. History of autonomic dysfunction, including amyloidosis, Parkinson's disease, autoimmune disease, spinal cord injury

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Migdal, MD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices) will be available for sharing.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing beginning 6 months after publication of findings from this study and ending 5 years after publication.
Access Criteria: Data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve the aims in the approved proposal. Requests to access the data should be directed to amigdal@emory.edu. To gain access, data requestors will need to sign a data access agreement

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital and Clinics, and Grady Health System in Atlanta, Georgia, USA. Participant enrollment began October 23, 2020 and all follow-up assessments were completed by February 8, 2022.
Period: Overall Study
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Started | 2 | 3
Completed | 1 | 0
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (10.5) | 54.7 (8.37) | 54.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: The hemoglobin A1c test result reflects average blood sugar level for the past two to three months. Specifically, the A1c test measures what percentage of hemoglobin is coated with sugar (glycated). The higher A1c level, the poorer blood sugar control and the higher risk of diabetes complications.
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: This analysis includes participants who attended the indicated study visit. One participant from the cryoablation plus lifestyle intervention group withdrew after the Month 6 visit. All three participants in the lifestyle intervention group were withdrawn or lost to follow up prior to the Month 3 visit.
Measure: Mean (Standard Deviation); unit: percent of glycated hemoglobin
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
percent of glycated hemoglobin
  Baseline | 8.35 (0.25) | 8.86 (0.40)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 8.75 (0.05) |
  Month 6: number analyzed (Participants) | 2 | 0
  Month 6 | 8.40 (0.20) |
  Month 12: number analyzed (Participants) | 1 | 0
  Month 12 | 9.30 (0.0) |

2. Primary Outcome: Insulin Resistance Score Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: Insulin resistance score HOMA-IR is computed with the formula: fasting plasma glucose (mmol/l) times fasting serum insulin (mU/l) divided by 22.5. Low HOMA-IR values indicate high insulin sensitivity, whereas high HOMA-IR values indicate low insulin sensitivity (insulin resistance).
Time Frame: Baseline, Month 3, Month 6, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (mmol/l X mU/l) / 22.5
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
(mmol/l X mU/l) / 22.5
  Baseline | 7.85 (1.75) | 4.70 (2.94)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 7.00 (1.00) |
  Month 6: number analyzed (Participants) | 2 | 0
  Month 6 | 10.70 (1.60) |
  Month 12: number analyzed (Participants) | 1 | 0
  Month 12 | 7.00 (0.0) |

3. Primary Outcome: Number of Deaths Among Recipients of the Cryoablation
Description: Mortality among recipients of the cryoablation was documented.
Time Frame: Up to Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention
Number analyzed (Participants) | 2
Participants | 0

4. Primary Outcome: Number of Adverse Events Related to the Cryoablation
Description: The count of procedure related complications, such as bleeding, infection, pneumothorax, hemothorax, pulmonary injury, complications of sedation, pain requiring hospital admission or treatment, dysphagia, gastroparesis, nausea and vomiting, and gastrointestinal ulceration was documented for the duration of the study.
Time Frame: Up to Month 12
Measure: Number; unit: related complications
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention
Number analyzed (Participants) | 2
related complications | 0

5. Secondary Outcome: Body Mass Index (BMI)
Description: Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters.
Time Frame: Baseline, Month 3, Month 6
Population: One participant from the cryoablation plus lifestyle intervention group attended the Month 6 study visit but did not complete all study activities for that visit. All three participants in the lifestyle intervention group were withdrawn or lost to follow up prior to the Month 3 visit.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
kg/m^2
  Baseline | 37.25 (1.55) | 33.26 (3.71)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 37.25 (0.25) |
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 39.5 (0.0) |

6. Secondary Outcome: Waist Circumference
Description: Waist circumference is a measurement taken around the abdomen at the level of the umbilicus (belly button). Waist circumference is measured in centimeters.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
cm
  Baseline | 121.3 (9.5) | 147.66 (58.39)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 117.5 (2.5) |
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 127 (0.0) |

7. Secondary Outcome: Waist-to-hip Ratio
Description: A waist-to-hip ratio of greater than 1.0 indicates a higher risk of developing heart disease. For women, a healthy waist-to-hip ratio is less than 0.85 while under 0.9 is a healthy ratio for men.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: waist cm/hip cm
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
waist cm/hip cm
  Baseline | 0.97 (0.02) | 1.06 (0.04)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 0.95 (0.05) |
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 1.0 (0.0) |

8. Secondary Outcome: Total Cholesterol
Description: A healthy level of total cholesterol is 125 - 200 mg/dL.
Time Frame: Baseline, Month 6
Population: This analysis includes participants who attended the indicated study visit. All three participants in the lifestyle intervention group were withdrawn or lost to follow up prior to the Month 3 visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
mg/dL
  Baseline | 198.00 (39.00) | 194.33 (39.19)
  Month 6: number analyzed (Participants) | 2 | 0
  Month 6 | 179.00 (42.00) |

9. Secondary Outcome: Low-Density Lipoprotein (LDL)
Description: A healthy level of LDL is less than 100 mg/dL.
Time Frame: Baseline, Month 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
mg/dL
  Baseline | 120.5 (30.5) | 121.33 (30.61)
  Month 6: number analyzed (Participants) | 2 | 0
  Month 6 | 102.0 (36.0) |

10. Secondary Outcome: Triglycerides
Description: A healthy level of triglycerides is less than 150 mg/dL.
Time Frame: Baseline, Month 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
mg/dL
  Baseline | 110 (16) | 151 (82)
  Month 6: number analyzed (Participants) | 2 | 0
  Month 6 | 85 (9) |

11. Secondary Outcome: Systolic Blood Pressure
Description: A normal systolic blood pressure level is less than 120 millimeters of mercury (mmHg).
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
mmHg
  Baseline | 127.00 (14.00) | 139.66 (8.17)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 112.50 (5.50) |
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 113.0 (0.0) |

12. Secondary Outcome: Diastolic Blood Pressure
Description: A normal diastolic blood pressure level is less than 80 mmHg.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
mmHg
  Baseline | 80.00 (2.00) | 80.66 (8.21)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 74.00 (0.00) |
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 80.00 (0.00) |

13. Secondary Outcome: Daily Caloric Intake
Description: Daily caloric intake is measured by 3-day food recall. Mean daily caloric intake is assessed as kilocalories (kcal) consumed per day.
Time Frame: Baseline, Month 3, Month 6
Population: The 3-day food recall diary was not completed by any study participants.
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Anti-hyperglycemic Medication Regimen
Description: Anti-hyperglycemic medications will be adjusted at visits under the direction of the endocrinologist, or as needed for clinically significant hypo- or hyperglycemic events. Changes in baseline medication regimen will be examined to determine if medication needs decrease or increase during the study.
Time Frame: Month 3, Month 6
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 0
Participants
  No change in dose from Baseline to Month 3 | 1 |
  Dose Increase from Baseline to Month 3 | 1 |
  No Change in Dose from Month 3 to Month 6 | 2 |

15. Secondary Outcome: Appetite Visual Analog Scale Score for Hunger
Description: The Appetite Visual Analog Scale includes 8 items which are scored on 100-mm visual analogue scales. The item for hunger asks participants how hungry they feel, where 0 = not at all and 100 = never been more hungry.
Time Frame: Baseline, Week 1, Month 1, Month 3, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
units on a scale
  Baseline | 98 (2) | 50 (37.96)
  Week 1 | 60.5 (35.5) | 60.5 (0.5)
  Month 1 | 26.5 (16.5) | 46 (3)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 34 (27) |
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 75 (0) |

16. Secondary Outcome: Appetite Visual Analog Scale Score for Satisfaction
Description: The Appetite Visual Analog Scale includes 8 items which are scored on 100-mm visual analogue scales. The item for satisfaction asks participants how satisfied they feel, where 0 = completely empty and 100 = cannot eat another bite.
Time Frame: Baseline, Week 1, Month 1, Month 3, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
units on a scale
  Baseline | 2.5 (2.5) | 19 (21.95)
  Week 1 | 37 (32) | 41.5 (10.5)
  Month 1 | 72 (19) | 41.5 (11.5)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 51 (20) |
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 35 (0) |

17. Secondary Outcome: Appetite Visual Analog Scale Score for Fullness
Description: The Appetite Visual Analog Scale includes 8 items which are scored on 100-mm visual analogue scales. The item for fullness asks participants how full they feel, where 0 = not full at all and 100 = totally full.
Time Frame: Baseline, Week 1, Month 1, Month 3, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
units on a scale
  Baseline | 2 (2) | 19.66 (21.45)
  Week 1 | 37.5 (33.5) | 28.5 (21.5)
  Month 1 | 77.5 (20.5) | 36 (21)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 53.5 (46.5) |
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 14 (0) |

18. Secondary Outcome: Appetite Visual Analog Scale Score for Eating Quantity
Description: The Appetite Visual Analog Scale includes 8 items which are scored on 100-mm visual analogue scales. The item for eating quantity asks participants how much they think they can eat, where 0 = nothing at all and 100 = a lot.
Time Frame: Baseline, Week 1, Month 1, Month 3, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
units on a scale
  Baseline | 74.5 (25.5) | 42.33 (13.88)
  Week 1 | 38 (11) | 52.5 (13.5)
  Month 1 | 35 (10) | 45 (20)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 31.5 (7.5) |
  Month 6: number analyzed (Participants) | 1 | 0
  Month 6 | 75 (0) |

19. Secondary Outcome: Appetite Visual Analog Scale Score for Desire for Certain Foods
Description: The Appetite Visual Analog Scale includes 8 items which are scored on 100-mm visual analogue scales. Four items of the questionnaire ask participants if they would like to eat something sweet, salty, savory, and fatty. Each item is scored as 0 = yes, very much and 100 = no, not at all.
Time Frame: Baseline, Week 1, Month 1, Month 3, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
units on a scale
  Baseline - Sweet | 23.5 (23.5) | 49.33 (40.83)
  Week 1 - Sweet | 37 (32) | 41.5 (10.5)
  Month 1 - Sweet | 75 (13) | 71 (9)
  Month 3 - Sweet: number analyzed (Participants) | 2 | 0
  Month 3 - Sweet | 42.5 (7.5) |
  Month 6 - Sweet: number analyzed (Participants) | 1 | 0
  Month 6 - Sweet | 47 (0) |
  Baseline - Salty | 23 (23) | 53.33 (31.75)
  Week 1 - Salty | 57.5 (11.5) | 57.5 (12.5)
  Month 1 - Salty | 32 (8) | 53 (13)
  Month 3 - Salty: number analyzed (Participants) | 2 | 0
  Month 3 - Salty | 46.5 (1.5) |
  Month 6 - Salty: number analyzed (Participants) | 1 | 0
  Month 6 - Salty | 53 (0) |
  Baseline - Savory | 11 (11) | 46 (36.80)
  Week 1 - Savory | 44 (22) | 61.5 (1.5)
  Month 1 - Savory | 71.5 (2.5) | 62.5 (11.5)
  Month 3 - Savory: number analyzed (Participants) | 2 | 0
  Month 3 - Savory | 43.5 (16.5) |
  Month 6 - Savory: number analyzed (Participants) | 1 | 0
  Month 6 - Savory | 25 (0) |
  Baseline - Fatty | 34.5 (34.5) | 60.66 (32.26)
  Week 1 - Fatty | 57 (12) | 38 (20)
  Month 1 - Fatty | 74.5 (1.5) | 60.5 (12.5)
  Month 3 - Fatty: number analyzed (Participants) | 2 | 0
  Month 3 - Fatty | 51.5 (6.5) |
  Month 6 - Fatty: number analyzed (Participants) | 1 | 0
  Month 6 - Fatty | 70 (0) |

20. Secondary Outcome: International Physical Activity Questionnaire (IPAQ) Score
Description: The IPAQ assesses physical activity during the past 7 days with 27 items. Based on the type, duration, and frequency of activity, respondents are categorized as having low activity, moderate activity, or high activity.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
Participants
  Baseline - Low activity | 0 | 1
  Baseline - Moderate activity | 0 | 2
  Baseline - High activity | 2 | 0
  Month 3 - Low activity: number analyzed (Participants) | 2 | 0
  Month 3 - Low activity | 1 |
  Month 3 - Moderate activity: number analyzed (Participants) | 2 | 0
  Month 3 - Moderate activity | 1 |
  Month 3 - High activity: number analyzed (Participants) | 2 | 0
  Month 3 - High activity | 0 |
  Month 6 - Low activity: number analyzed (Participants) | 2 | 0
  Month 6 - Low activity | 2 |
  Month 6 - Moderate activity: number analyzed (Participants) | 2 | 0
  Month 6 - Moderate activity | 0 |
  Month 6 - High activity: number analyzed (Participants) | 2 | 0
  Month 6 - High activity | 0 |

21. Secondary Outcome: Fasting Glucose Level
Description: A normal fasting blood sugar level is 99 mg/dL or lower, glucose levels of 100 - 125 mg/dL indicates prediabetes, and levels of 126 mg/dL and higher indicates diabetes.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
mg/dL
  Baseline | 197 (25) | 166.33 (4.64)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 186.5 (28.5) |
  Month 6: number analyzed (Participants) | 2 | 0
  Month 6 | 151.5 (4.5) |

22. Secondary Outcome: Fasting Insulin Level
Description: A normal fasting insulin level for the Emory Healthcare Laboratory is 1.9 to 23.0 milli-international units per liter (mIU/L). High levels of fasting insulin are associated with obesity and early stage type 2 diabetes (T2D). Type 1 diabetes and advanced T2D are associated with low levels of insulin.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
Number analyzed (Participants) | 2 | 3
mIU/L
  Baseline | 15.9 (1.6) | 11.6 (7.65)
  Month 3: number analyzed (Participants) | 2 | 0
  Month 3 | 16.5 (4.1) |
  Month 6: number analyzed (Participants) | 2 | 0
  Month 6 | 18.65 (6.35) |

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time individuals gave consent to participate in the study and continued through the 12 Month study visit.
Arm/Group | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention | Lifestyle Intervention Only
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoablation of the Vagus Nerve Plus Lifestyle Intervention (N=2) | Lifestyle Intervention Only (N=3)
Right upper quadrant abdominal pain (Gastrointestinal disorders) | 1 | 0
Dizziness (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT04276051/Prot_SAP_000.pdf